CLINICAL TRIAL: NCT01820962
Title: Concentrated Citrate Locking to Reduce the Incidence of Central Venous Catheter-related Infections and Thrombosis: a Randomized Phase III Study in a Hematological Patient Population
Brief Title: Concentrated Citrate Locking to Reduce the Incidence of CVC-related Complications in Hematological Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Because the inclusion rate was lower than expected.
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Dirinco B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MEC06-2-003
Record Dates: First submitted 2013-03-12; First posted 2013-03-29 (Estimated); Last update posted 2013-03-29 (Estimated); Status verified 2013-03

CONDITIONS: Hematological Malignancies; Bacteremia; Thrombosis
Keywords: hematological patients; central venous catheters; catheter related thrombosis; catheter related infections; concentrated citrate
MeSH Terms: conditions — Hematologic Neoplasms; Bacteremia; Thrombosis; Catheter-Related Infections | interventions — Heparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A: heparin (Heparin LEO) (Active Comparator): After each use, the central venous catheter lumen will be flushed with 10 ml 0.9% NaCl and then locked with heparin 5000 IU/ml(standard treatment)using a volume exactly equivalent to the internal volume noted on each catheter.
  Interventions: Procedure: heparin
- B: concentrated citrate (Citralock) (Experimental): locking the central venous catheter with concentrated citrate after each use
  Interventions: Procedure: concentrated citrate

INTERVENTIONS:
Procedure: heparin — when not in use CVCs are locked with heparin
  Arms: A: heparin (Heparin LEO)
Procedure: concentrated citrate — when not in use the CVC is locked with concentrated citrate
  Arms: B: concentrated citrate (Citralock)

SUMMARY:
Patients with a hematological malignancy who are undergoing intensive chemotherapy need a central venous catheter (CVC)during their treatment. CVCs are locked with heparin when they are not used.

The purpose of this study is to determine whether concentrated citrate locking, compared to heparin, reduces the incidence of central venous catheter-related thrombosis and infections in patients with hematological malignancies undergoing intensive chemotherapy.

DETAILED DESCRIPTION:
Central venous catheter (CVC)-related thrombosis and infections are frequently occurring complications and may cause significant morbidity in patients with hematological malignancies. Interventions to decrease fibrin deposition have the potential to reduce CVC-related thrombosis and infections.

At present heparin is most often used as locking solution for central venous catheters in hematological patients despite a lack of evidence regarding the efficacy and safety. Trisodium citrate (TSC) had been shown to be an effective antimicrobial catheter locking in hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* patients with hematological malignancies who were going to receive a CVC for intensive chemotherapy including patients for stem cell transplantation
* written informed consent
* 18 years or older

Exclusion Criteria:

* the presence of a central venous catheter at admission
* history of central venous catheter related thrombosis or infection
* indication for anticoagulant treatment or prophylaxis
* patients with totally implanted catheters
* catheters impregnated with antimicrobial agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2006-07; Primary Completion 2010-12 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
central venous catheter-related thrombosis | weekly from date of randomization until removal of the central venous catheter, up to one year
  Patients will be followed from insertion of the central venous catheter till removal of the central venous catheter, an expected average of 30 days. The central venous catheter is seen daily and checked for thrombosis and infections when the patient is admitted on the ward. Discharged patients are seen at least weekly on the outpatients clinic and their central venous catheter is checked for thrombosis and infections. A standard ultrasound is made 30 days after insertion and within 24 hours after removal of the central venous catheter.
central venous catheter-related infections | weekly from date of randomization untill the removal of the central venous catheter; up to one year

SECONDARY OUTCOMES:
premature removal of the catheter | weekly from date of randomization untill removal of the central venous catheter; up to one year
failure to aspirate blood | weekly from date of randomization untill the removal of the central venous catheter; up to one year
hypocalcemic symptoms | weekly from dateof randomization untill the removal of the central venous catheter; up to one year
severe bleeding | weekly from date of randomization untill the removal of the central venous catheter; up to one year

CONTACTS AND LOCATIONS:
Overall Officials: Harry Schouten, MD, Principal Investigator — Maastricht University Medical Centre
Locations (2):
- Netherlands (2):
  - Atrium Medical Center Parkstad Heerlen, Heerlen
  - Maastricht University Medical Center, Maastricht

REFERENCES:
- [Background] Boersma RS, Jie KS, Verbon A, van Pampus EC, Schouten HC. Thrombotic and infectious complications of central venous catheters in patients with hematological malignancies. Ann Oncol. 2008 Mar;19(3):433-42. doi: 10.1093/annonc/mdm350. Epub 2007 Oct 24. PMID 17962211
- [Background] Raad I, Hanna H, Maki D. Intravascular catheter-related infections: advances in diagnosis, prevention, and management. Lancet Infect Dis. 2007 Oct;7(10):645-57. doi: 10.1016/S1473-3099(07)70235-9. PMID 17897607
- [Background] Weijmer MC, van den Dorpel MA, Van de Ven PJ, ter Wee PM, van Geelen JA, Groeneveld JO, van Jaarsveld BC, Koopmans MG, le Poole CY, Schrander-Van der Meer AM, Siegert CE, Stas KJ; CITRATE Study Group. Randomized, clinical trial comparison of trisodium citrate 30% and heparin as catheter-locking solution in hemodialysis patients. J Am Soc Nephrol. 2005 Sep;16(9):2769-77. doi: 10.1681/ASN.2004100870. Epub 2005 Jul 20. PMID 16033861